CLINICAL TRIAL: NCT03074201
Title: Prospective Evaluation of the Ability of Spyglass Cholangioscopy to Facilitate Radiation Free ERCP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: Boston Scientific Corporation (Industry)
Responsible Party: Principal Investigator, Subhas Banerjee, Associate Professor of Medicine, Stanford University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: 32194
Record Dates: First submitted 2017-02-23; First posted 2017-03-08 (Actual); Last update posted 2018-09-11 (Actual); Status verified 2018-09

CONDITIONS: Choledocholithiasis; Biliary Obstruction
Keywords: ERCP, choledocholithiasis, cholangioscopy
MeSH Terms: conditions — Choledocholithiasis

STUDY DESIGN:
Intervention Model Description: Prospective feasibility study to evaluate potential for cholangioscopy to facilitate radiation-free ERCP.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Cholangioscopy (Experimental): Participants in this arm undergo radiation-free ERCP facilitated by cholangioscopy
  Interventions: Procedure: Cholangioscopy; Device: Spyglass DS Cholangioscope

INTERVENTIONS:
Procedure: Cholangioscopy — Cholangioscopy used instead of fluoroscopy-based ERCP to facilitate clearance of bile duct stones.
Device: Spyglass DS Cholangioscope — Cholangioscopy used instead of fluoroscopy-based ERCP to facilitate clearance of bile duct stones.

SUMMARY:
Prospective Evaluation of the Ability of Spyglass Cholangioscopy to Facilitate Radiation Free ERCP for non-complex bile duct stone disease.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 and above
2. Non-complex biliary stone disease involving stones in the common bile or common hepatic duct.
3. Patient has undergone non-invasive imaging (abdo US, MRCP etc) which clearly delineates bile duct diameter and suggests non complex biliary stone disease.
4. Willing and able to comply with the study procedures and provide written informed consent to participate in the study.

Exclusion Criteria:

1. Age <18
2. Potentially vulnerable subjects including, homeless people, pregnant females, employees and students.
3. Participation in another related investigational study that could affect the results of this study within the previous 30 days
4. Complex biliary stone disease cases with unusual location of the stones (intra hepatic, cystic duct, stone proximal to bile duct stricture)
5. Known bile duct infection (cholangitis defined as ongoing fevers on the day of the ERCP procedure or purulence evident at the ampulla or bile duct on cannulation/sphincterotomy. If clear bile is aspirated during the study procedure, we will proceed according to study procedures. If purulence is detected upon aspiration of bile during the procedure, patient will be excluded from the study and undergo standard radiation-based ERCP rather than cholangioscopy.)

5) Complex post-surgical anatomy e.g. Billroth type II anatomy, Roux-en-Y-gastrojejunostomy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2015-10-01 (Actual); Primary Completion 2017-05-20 (Actual); Study Completion 2017-05-20 (Actual)

PRIMARY OUTCOMES:
Stone clearance | During the cholangioscopy procedure
  Successful clearance of stones from the bile duct using cholangioscopy

SECONDARY OUTCOMES:
Procedure Duration | 5 minutes to 2.5 hours anticipated time frame
  Duration of procedure

OTHER OUTCOMES:
Adverse Events | up to 30 weeks post-procedure
  Evaluation of adverse events following the procedure

CONTACTS AND LOCATIONS:
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States

REFERENCES:
- [Derived] Barakat MT, Girotra M, Choudhary A, Huang RJ, Sethi S, Banerjee S. A prospective evaluation of radiation-free direct solitary cholangioscopy for the management of choledocholithiasis. Gastrointest Endosc. 2018 Feb;87(2):584-589.e1. doi: 10.1016/j.gie.2017.07.042. Epub 2017 Aug 7. PMID 28797911